CLINICAL TRIAL: NCT02597062
Title: A Single Arm Phase II Study of High-Dose Weekly Carfilzomib Plus Cyclophosphamide and Dexamethasone in the Treatment of Relapsed Multiple Myeloma After 1-3 Prior Therapies
Brief Title: High-Dose Weekly Carfilzomib Plus Cyclophosphamide and Dexamethasone in the Treatment of Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Amgen (Industry); Canadian Myeloma Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYX1; MCRN003 (Other: MCRN)
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2022-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carfilzomib plus cyclophosphamide plus dexamethasone (Experimental): 20 mg/m2 day 1 of first cycle then escalated to 70 mg/m2 for all subsequent doses) given on days 1, 8, and 15 of a 28 day cycle plus weekly oral dexamethasone (< 70 years, 40 mg; ≥ 70 years 20mg) and cyclophosphamide 300 mg/m2 capped at 500 mg
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib
Drug: Cyclophosphamide
Drug: Dexamethasone

SUMMARY:
The purpose of this study is to find out what effects carfilzomib has on relapsed multiple myeloma when administered in combination with cyclophosphamide and dexamethasone.

DETAILED DESCRIPTION:
Multiple Myeloma is a cancer that affects the bone marrow where the cells in our blood system are formed. This includes the white cells, red cells, platelets and lymphoid cells. In multiple myeloma the plasma cell (one of the lymphoid cells) starts to reproduce out of control. This results in crowding of the bone marrow with abnormal production of all the cells and a malfunction of the plasma cells. They can also cause damage to the normal bone resulting in pain, fractures and other complications.

The standard or usual treatments for your disease are lenalidomide (an immunomodulatory drug) or bortezomib (a proteasome inhibitor) based treatments.

Carfilzomib is a new type of proteasome inhibitor that is approved for the treatment of relapsed multiple myeloma in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed symptomatic multiple myeloma as per the International Myeloma Working group criteria [Palumbo 2009].
* Measurable disease, as defined by one or more of the following (assessed within 21 days prior to registration):

  * Serum M-protein ≥ 5 g/L (0.5g/dL)
  * Urine Bence-Jones protein ≥ 200 mg/24 hours
  * Involved serum free light chain (FLC) measurement ≥ 100 mg/L (10 mg/dL), provided serum FLC ratio is abnormal (abnormal if FLC ratio is <0.26 or >1.65)
  * Biopsy proven plasmacytoma
  * For IgA patients whose disease can only be reliably measured by serum quantitative immunoglobulin (qIgA) ≥ 750 mg/dL (0.75 g/dL)
* Prior treatment with at least one, but no more than three, regimens for multiple myeloma
* Documented relapse or progressive disease on or after any regimen (subjects refractory to the most recent line of therapy are eligible except those who are refractory to bortezomib and cyclophosphamide as described in exclusion criteria 1.
* Achieved a response to at least one prior regimen (defined as ≥ 25% decrease in M-protein)
* Age ≥ 18 years.
* Life expectancy ≥ 3 months.
* ECOG performance status 0-2.
* Laboratory Requirements (must be done within 21 days of registration):
* Hematology:

  * Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L
  * Hemoglobin ≥ 8 g/dL (80 g/L) (subjects may be receiving red blood cell (RBC) transfusions in accordance with institutional guidelines)
  * Platelet count ≥ 50 × 10^9/L, independent of platelet transfusions for 7 days. (≥ 30 × 10^9/L if myeloma involvement in the bone marrow is ≥ 50%)
* Biochemistry:

  * ALT ≤ 3.5 x UNL
  * Serum direct bilirubin ≤ 2 mg/dL (34 μmol/L) (only required if total bilirubin ≥ 2mg/dL (34μmol/L)
  * Creatinine clearance (CrCl) ≥ 30 mL/minute (Crockcroft and Gault formula) and not on dialysis.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre.
* In accordance with CRO policy, protocol treatment is to begin within 2 working days of patient registration.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method.

Exclusion Criteria:

* Refractory to any proteasome inhibitor therapy (bortezomib, ixazomib, etc.) Refractory disease is defined as failure to respond to the proteasome inhibitor, initial response followed by progression while on a proteasome inhibitor, or relapse within 60 days of stopping proteasome inhibitor therapy.
* Prior carfilzomib treatment.
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Waldenström's macroglobulinemia or IgM myeloma
* Current or previous Plasma cell leukemia defined as (> 2.0 × 10^9/L circulating plasma cells by standard differential)
* Chemotherapy or investigational agent within 3 weeks prior to registration or antibody therapy within 6 weeks prior to registration
* Radiotherapy to multiple sites within 28 days prior to registration; localized radiotherapy to a single site within 7 days prior to registration
* Plasmapheresisis within 14 days of registration.
* Pregnant or lactating females.
* Major surgery within 21 days prior to registration.
* Active, uncontrolled bacterial, fungal, or viral infection.
* Concurrent amyloidosis
* Known human immunodeficiency virus infection.
* Active hepatitis B or C infection.
* Myocardial infarction within 4 months prior to registration, NYHA Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or grade 3 conduction system abnormalities unless subject has a pacemaker.
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to registration.
* Other malignancy, including MDS, within the past 3 years with the exception of adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; carcinoma in situ of the cervix or breast; prostate cancer of Gleason Score 6 or less with stable prostate-specific antigen levels; or cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumours of the adrenal or pancreas.
* Significant neuropathy (≥ grade 3, or grade 2 with pain) within 14 days prior to registration.
* Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib).
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment.
* Ongoing graft-versus-host disease.
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to registration.
* Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Venner, Study Chair — Cross Cancer Institute, Edmonton Alberta Canada
Locations (9):
- Canada (9):
  - Cross Cancer Institute, Edmonton, Alberta
  - Regional Health Authority B, Zone 2, Saint John, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - CIUSSS de l'Est-de-I'lle-de-Montreal, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Venner CP, LeBlanc R, Sandhu I, White D, Belch AR, Reece DE, Chen C, Dolan S, Lalancette M, Louzada M, Kew A, McCurdy A, Monteith B, Reiman T, McDonald G, Sherry M, Gul E, Chen BE, Hay AE. Weekly carfilzomib plus cyclophosphamide and dexamethasone in the treatment of relapsed/refractory multiple myeloma: Final results from the MCRN-003/MYX.1 single arm phase II trial. Am J Hematol. 2021 May 1;96(5):552-560. doi: 10.1002/ajh.26147. PMID 33650179
- [Derived] Monteith BE, Venner CP, Reece DE, Kew AK, Lalancette M, Garland JS, Shepherd LE, Pater JL, Hay AE. Drug-induced Thrombotic Microangiopathy with Concurrent Proteasome Inhibitor Use in the Treatment of Multiple Myeloma: A Case Series and Review of the Literature. Clin Lymphoma Myeloma Leuk. 2020 Nov;20(11):e791-e800. doi: 10.1016/j.clml.2020.04.014. Epub 2020 Apr 30. PMID 32807717

RESULTS

PARTICIPANT FLOW:
Groups:
- Carfilzomib Plus Cyclophosphamide Plus Dexamethasone: 20 mg/m2 day 1 of first cycle then escalated to 70 mg/m2 for all subsequent doses) given on days 1, 8, and 15 of a 28 day cycle plus weekly oral dexamethasone (< 70 years, 40 mg; ≥ 70 years 20mg) and cyclophosphamide 300 mg/m2 capped at 500 mg
  Carfilzomib
  Cyclophosphamide
  Dexamethasone
Period: Overall Study
Arm/Group | Carfilzomib Plus Cyclophosphamide Plus Dexamethasone
Started | 76
Completed | 75
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Population: All eligible and treated patients
Arm/Group | Carfilzomib Plus Cyclophosphamide Plus Dexamethasone
Number analyzed (Participants) | 75
Age, Continuous [Median (Full Range); unit: years] | 66.0 [44.0 to 82.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 68
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Canada | 75

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate After 4 Cycles
Description: Response rate to protocol treatment after 4 cycles is define by stringent complete response, complete response, partial response, very good partial response, minimal response.
  Complete response: Negative immunofixation on the serum and urine and Disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow biopsy Stringent complete response: Complete response plus Absence of clonal cells in bone marrow d by immunohistochemistry or immunofluorescence Very good partial response: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein with urine M-protein level <100 mg/24 hours.
  Partial response: ≥50% reduction in serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours Minimal response: 25-49% reduction in serum M-protein, and 50-89% reduction in 24-hour urinary M-protein, if ≥ 200 mg/24 hours at baseline
Time Frame: 4 months
Population: All eligible patients how have received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Plus Cyclophosphamide Plus Dexamethasone
Number analyzed (Participants) | 75
Participants
  stringent complete response | 4
  complete response | 3
  very good partial response | 32
  partial response | 21
  minimal response | 1
  no response | 14

2. Secondary Outcome: Progression-free Survival
Description: Median time to progression or death assessed by biochemistry, radiology and immunology tests will be reported. Progression is evaluated in this study using the International Myeloma Working Group Uniform Response Criteria (IMWG-URC) with any one or more of the following:
  1. Increase of ≥ 25% from lowest response value in: Serum M-component and/or Urine M-component and/or Only in patients without measurable serum and urine M-protein levels; the difference between involved and uninvolved FLC levels or Bone marrow plasma cell percentages.
  2. Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
  3. Development of hypercalcemia (corrected serum calcium > 11.5 mg/dL (0.115 g/L) or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: 3 years
Population: All treated patients were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib Plus Cyclophosphamide Plus Dexamethasone
Number analyzed (Participants) | 75
months | 17.15 [13.57 to 21.49]

3. Secondary Outcome: Overall Survival
Description: Median time to death in months will be reported
Time Frame: 3 years
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib Plus Cyclophosphamide Plus Dexamethasone
Number analyzed (Participants) | 75
months | 27.43 [22.05 to 33.8]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Carfilzomib Plus Cyclophosphamide Plus Dexamethasone
All-Cause Mortality (participants affected / at risk) | 31/75
Serious Adverse Events (participants affected / at risk) | 39/75
Other Adverse Events (participants affected / at risk) | 28/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib Plus Cyclophosphamide Plus Dexamethasone (N=75)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Other blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2
Heart failure (Cardiac disorders) | 2
Mitral valve disease (Cardiac disorders) | 1
Right ventricular dysfunction (Cardiac disorders) | 1
Death NOS (General disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 4
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Abdominal infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 14
Other infections and infestations (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Upper respiratory infection (Infections and infestations) | 3
Ankle fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Other neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ischemia cerebrovascular (Nervous system disorders) | 1
Other nervous system disorders (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Other vascular disorders (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib Plus Cyclophosphamide Plus Dexamethasone (N=75)
Fatigue (General disorders) | 12
Lung infection (Infections and infestations) | 15
Sepsis (Infections and infestations) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT02597062/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT02597062/SAP_001.pdf